CLINICAL TRIAL: NCT00888238
Title: A Randomized Clinical Trial to Evaluate Glucose-Dependent Insulinotropic Effects of a Single Dose of a DPP-4 Inhibitor in Lean Healthy Males
Brief Title: A Method to Evaluate Glucose-Dependent Insulin Secretion in Healthy Males (MK-0431-179)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: 0431-179; 2009_584 (Other: Merck Registration Number); CTRI/2009/091/000457 (Registry Identifier: CTRI)
Record Dates: First submitted 2009-04-24; First posted 2009-04-27 (Estimated); Results first posted 2010-08-03 (Estimated); Last update posted 2018-06-26 (Actual); Status verified 2018-03

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Sitagliptin/Sitagliptin/Placebo (Experimental): Sitagliptin in 2 of 3 treatment periods and Placebo in 1 of 3 treatment periods
  Interventions: Drug: sitagliptin; Drug: Comparator: Placebo
- Sitagliptin/Placebo/Sitaglipitin (Experimental): Sitagliptin in 2 of 3 treatment periods and Placebo in 1 of 3 treatment periods
  Interventions: Drug: sitagliptin; Drug: Comparator: Placebo
- Placebo/Sitagliptin/Sitagliptin (Experimental): Sitagliptin in 2 of 3 treatment periods and Placebo in 1 of 3 treatment periods
  Interventions: Drug: sitagliptin; Drug: Comparator: Placebo

INTERVENTIONS:
Drug: sitagliptin — Single oral dose of sitagliptin 100 mg (2 x 50 mg) tablets followed by the hyperglycemic clamp procedure and meal tolerance test.
  Other Names: sitagliptin phosphate; MK0431
Drug: Comparator: Placebo — Single oral dose of 2 tablets placebo to sitagliptin followed by the hyperglycemic clamp procedure and meal tolerance test.

SUMMARY:
This study will evaluate the effect of a single dose of sitagliptin on glucose dependent insulin secretion using a meal tolerance test (MTT) during a hyperglycemic clamp (HCG) procedure.

ELIGIBILITY:
Inclusion Criteria:

* Subject is an Asian Indian male between 18 to 45 years of age
* Subject is in good health
* Subject is a nonsmoker or has not used nicotine-containing products for six months
* Subject is willing to avoid strenuous activity

Exclusion Criteria:

* Subject has a history of stroke, seizures, or major neurological disorders
* Subject has irritable bowel disease or recurrent nausea, vomiting, diarrhea, or abdominal pain
* Subject has a history of high blood pressure requiring treatment
* Subject has history of cancer
* Subject has a history of diabetes

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2009-05-12 (Actual); Primary Completion 2009-06-10 (Actual); Study Completion 2009-07-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Shankar SS, Shankar RR, Mixson LA, Miller DL, Steinberg HO, Beals CR, Kelley DE. Insulin secretory effect of sitagliptin: assessment with a hyperglycemic clamp combined with a meal challenge. Am J Physiol Endocrinol Metab. 2018 Apr 1;314(4):E406-E412. doi: 10.1152/ajpendo.00238.2017. Epub 2017 Nov 14. PMID 29138226

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited at Veeda Clinical Research Pvt. Ltd. in May 2009.
  First Patient Screened: 20-May-2009.
  Last Patient, Last Visit: 21-Jul-2009.
  1 site
Pre-assignment Details: Subjects screened over a 1 week period.
Groups:
- Sitagliptin / Sitagliptin / Placebo: Single oral dose Sitagliptin 100 mg (administered as 2 X 50 mg tablet) / Single oral dose Sitagliptin 100 mg (administered as 2 X 50 mg tablet) / Matching Placebo
- Sitagliptin / Placebo / Sitagliptin: Single oral dose Sitagliptin 100 mg (administered as 2 X 50 mg tablet) / Matching Placebo / Single oral dose Sitagliptin 100 mg (administered as 2 X 50 mg tablet)
- Placebo / Sitagliptin / Sitagliptin: Matching Placebo / Single oral dose Sitagliptin 100 mg (administered as 2 X 50 mg tablet) / Single oral dose Sitagliptin 100 mg (administered as 2 X 50 mg tablet)
Period: First Period of Treatment Intervention
Arm/Group | Sitagliptin / Sitagliptin / Placebo | Sitagliptin / Placebo / Sitagliptin | Placebo / Sitagliptin / Sitagliptin
Started | 4 | 4 | 4
Completed | 4 | 4 | 4
Not Completed | 0 | 0 | 0
Period: Washout Period After Period 1
Arm/Group | Sitagliptin / Sitagliptin / Placebo | Sitagliptin / Placebo / Sitagliptin | Placebo / Sitagliptin / Sitagliptin
Started | 4 | 4 | 4
Completed | 4 | 4 | 4
Not Completed | 0 | 0 | 0
Period: Second Period of Treatment Intervention
Arm/Group | Sitagliptin / Sitagliptin / Placebo | Sitagliptin / Placebo / Sitagliptin | Placebo / Sitagliptin / Sitagliptin
Started | 4 | 4 | 4
Completed | 4 | 4 | 4
Not Completed | 0 | 0 | 0
Period: Washout Period After Period 2
Arm/Group | Sitagliptin / Sitagliptin / Placebo | Sitagliptin / Placebo / Sitagliptin | Placebo / Sitagliptin / Sitagliptin
Started | 4 | 4 | 4
Completed | 4 | 4 | 3
Not Completed | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 1
Period: Third Period of Treatment Intervention
Arm/Group | Sitagliptin / Sitagliptin / Placebo | Sitagliptin / Placebo / Sitagliptin | Placebo / Sitagliptin / Sitagliptin
Started | 4 | 4 | 3
Completed | 4 | 4 | 3
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Patients: All Randomized patients
Arm/Group | All Patients
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.8 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 12
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 20.5 (1.3)

OUTCOME MEASURES:

1. Primary Outcome: Insulin Secretion Rate (ISR) During 190 - 340 Minutes Post-dose
Description: ISR was estimated by the deconvolution of peripheral C-peptide concentrations using a 2-compartment model that utilizes population C-peptide kinetic parameters.
Time Frame: 190 minutes to 340 minutes
Population: All subjects who completed a hyperglycemic clamp in each period were included in the analysis.
Measure: Least Squares Mean (Standard Deviation); unit: ng/min
Groups:
- Sitagliptin 100 mg: 11 subjects received a single-dose of sitagliptin 100 mg in 2 periods; 1 subject received a single dose of sitagliptin 100 mg in 1 period only.
- Placebo: 12 subjects received a single-dose of placebo in 1 period.
Arm/Group | Sitagliptin 100 mg | Placebo
Number analyzed (Participants) | 12 | 12
ng/min | 9.73 (2.72) | 8.03 (2.58)
Statistical Analysis 1: Comparison: Sitagliptin 100 mg vs Placebo; Test type: Superiority or Other; p < 0.001, ANOVA; Least Squares Mean = 1.70, 90% CI [1.47 to 1.93]

2. Secondary Outcome: Glucose Infusion Rate (GIR) During 190 - 340 Minutes Post-dose
Description: Glucose Infusion Rate required to maintain the target glucose level of 160 milligrams / deciliter (mg/dL) ; GIR was normalized to subject's body weight (kg).
Time Frame: 190 minutes to 340 minutes
Population: All subjects who completed a hyperglycemic clamp in each period were included in the analysis.
Measure: Least Squares Mean (Standard Deviation); unit: mg / kg / min
Arm/Group | Sitagliptin 100 mg | Placebo
Number analyzed (Participants) | 12 | 12
mg / kg / min | 15.0 (2.6) | 13.7 (2.3)
Statistical Analysis 1: Comparison: Sitagliptin 100 mg vs Placebo; Test type: Superiority or Other; p < 0.001, ANOVA; Least Squares Mean = 1.30, 90% CI [1.08 to 1.52]

ADVERSE EVENTS:
Time Frame: Adverse experiences were collected from the time the consent was signed through the 14 day follow up period, after all treatment periods were completed.
Description: Subjects were queried at each visit for any adverse experiences since the previous visit.
Arm/Group | Sitagliptin 100 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 1/12 | 0/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sitagliptin 100 mg (N=12) | Placebo (N=12)
Blister (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.